CLINICAL TRIAL: NCT02869932
Title: Prospective Study of the Phenotypic Expression of Cystic Fibrosis (CF) Screened Positive Newborns With an Atypical Form of CF (DPAM)
Acronym: DPAM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Vaincre la Mucoviscidose (Other); French society of cystic fibrosis (Unknown); AFDPHE : newborn screening of the French Society of Cystic Fibrosis (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: P101003
Record Dates: First submitted 2015-01-09; First posted 2016-08-17 (Estimated); Last update posted 2023-02-06 (Actual); Status verified 2016-08

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Atypical and classic cystic fibrosis (Other): Lung CT scan without injection
  Interventions: Radiation: Lung CT scan

INTERVENTIONS:
Radiation: Lung CT scan — Lung CT scan without injection

SUMMARY:
The strategy of neonatal screening for Cystic Fibrosis in France relies on Immuno Reactive Trypsinogen (IRT) at day 3/DNA analysis with a CF Elucigen 30 mutations kit/ IRT safety-net at day 21. This strategy has significantly improved the performance of CF neonatal screening (NNS) in terms of positive predictive value and sensitivity but revealed new difficulties. Up to 85-90% of CF patients detected through the NNS program has a classical CF form with a positive sweat test and 2, 1 or no CF causing mutations but the remainder has either 2 CFTR mutations with at least one non-CF causing mutation and a sweat test <60mmol/L or 1, 0 CFTR mutation and an intermediate sweat test value ≥ 30 et < 60mmol/L raising a diagnosis and prognosis dilemma. Meanwhile the vast majority of these cohorts will remain asymptomatic over time, some will develop symptoms prompting clinicians to maintain a rigorous surveillance for the entire atypical cohort, whose modalities vary a lot among centers and countries.

This prospective multicenter study with a standardized assessment of a matched cohort with "atypical" CF versus "classical" CF from 6 years of age (60-65 cases in each cohort) is aimed at evaluating pulmonary and nutritional status to, better define the best monitoring follow-up, therapeutic management and familial genetic counseling.

DETAILED DESCRIPTION:
The strategy of neonatal screening for Cystic Fibrosis in France relies on Immuno Reactive Trypsinogen (IRT) at day 3/DNA analysis with a CF Elucigen 30 mutations kit/ IRT safety-net at day 21. This strategy has significantly improved the performance of CF neonatal screening (NNS) in terms of positive predictive value and sensitivity but revealed new difficulties. Up to 85-90% of CF patients detected through the NNS program has a classical CF form with a positive sweat test and 2, 1 or no CF causing mutations but the remainder has either 2 CFTR mutations with at least one non-CF causing mutation and a sweat test <60mmol/L or 1, 0 CFTR mutation and an intermediate sweat test value ≥ 30 et < 60mmol/L raising a diagnosis and prognosis dilemma. Meanwhile the vast majority of these cohorts will remain asymptomatic over time, some will develop symptoms prompting clinicians to maintain a rigorous surveillance for the entire atypical cohort, whose modalities vary a lot among centers and countries.

This prospective multicenter study with a standardized assessment of a matched cohort with "atypical" CF versus "classical" CF from 6 years of age (60-65 cases in each cohort) is aimed at evaluating pulmonary and nutritional status to, better define the best monitoring follow-up, therapeutic management and familial genetic counseling.

ELIGIBILITY:
Inclusion Criteria:

* Atypical CF cohort: children identified trough newborn screening on a hypertrypsinemia, who are older than 6 years of age at the time of inclusion and who carry a) 2 CFTR gene mutations of the CF30 kit with at least one R117H whatever the value of the sweat test or b) 2 CFTR gene mutations of the CF30 kit with a sweat test chloride < 60mmol/L or c) 1 or 0 mutation in the CF30 kit with a sweat test ≥ 30 and <60mmol/L and identification of additional mutations by comprehensive screening of the gene
* Classical CF cohort: children identified by newborn screening on a hypertrypsinemia, who are matched with an Atypical CF by age and sex if possible and who were diagnosed with a classical CF based on a sweat test > 60 mmol/ L with 0, 1 or 2 CF causing gene mutations.

Exclusion Criteria:

* • Drugs such as CFTR modulators interfering with the phenotypic expression of the disease.

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 130 (Actual)
Dates: Start 2012-03; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Comparison of Score Brody 2 (0 to 270) between the atypical and classical CF cohorts | 1 day
  Score Brody 2 (0 to 270) mesured by Lung CT scan without injection

SECONDARY OUTCOMES:
Comparison of Wisconsin and Brasfield scores between the atypical and classical CF cohorts | 1 day
  Wisconsin and Brasfield scores will be mesured by Chest X-ray

CONTACTS AND LOCATIONS:
Locations (1):
- Robert Debre Hospital - Assistance Puplique - Hôpitaux de Paris, Paris, France

REFERENCES:
- [Result] Munck A, Bourmaud A, Bellon G, Picq P, Farrell PM; DPAM Study Group. Phenotype of children with inconclusive cystic fibrosis diagnosis after newborn screening. Pediatr Pulmonol. 2020 Apr;55(4):918-928. doi: 10.1002/ppul.24634. Epub 2020 Jan 9. PMID 31916691